CLINICAL TRIAL: NCT04578314
Title: RELATE - A Randomized Controlled Trial of a Cognitive Behavioural Module for Distressing Auditory Verbal Hallucinations
Brief Title: RELATE - Efficacy and Feasibility of a Cognitive Behavioural Module for Distressing Auditory Verbal Hallucinations
Acronym: RELATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Collaborators: University of Leipzig (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Jacobs University Bremen gGmbH (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Matthias Pillny, Trial Manager, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 419676143
Record Dates: First submitted 2020-09-18; First posted 2020-10-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Verbal Auditory Hallucination; Psychotic Disorders; Psychosis; Schizophrenia
Keywords: Relating therapy
MeSH Terms: conditions — Hallucinations; Psychotic Disorders; Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, parallel-group, two-armed, multicentre, open trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relating module + Treatment as usual (Experimental): Participants in this arm will receive 16 weekly sessions with Relating Therapy (RT) over 5 months in addition to their treatment as usual.
  Interventions: Behavioral: Relating Therapy; Other: Treatment as usual
- Treatment as usual (Active Comparator): Treatment as usual will include medication management, supportive brief counselling sessions and various types of psychosocial (e.g. social work guided support, peer support) and monitoring provided by Mental Health Services, with individual and family psychological therapies offered occasionally. Individual therapies may include Cognitive Behavior Therapy or psychodynamic interventions.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Relating Therapy — Relating Therapy (RT) is a symptom-specific behaviourally oriented intervention that targets interpersonal relating as a key mechanism associated with auditory hallucination distress. The aim is that patients learn to relate more assertively within the difficult relationships they have with both the auditory hallucinations and other people. The RT will follow a treatment manual consisting of three phases: 1. Socialization to relating therapy and its implications; 2. Exploration of themes within the relational history of the participant and their experience of relationships with AH, and interpersonal relating within the family and social environment (identifying any prominent themes, such as abuse, disempowerment, or rivalry); 3. Exploration and development of assertive approaches to relating to AH and other people.
  Arms: Relating module + Treatment as usual
Other: Treatment as usual — TAU will include medication management, supportive brief counselling sessions and various types of psychosocial (e.g. social work guided support, peer support) and monitoring provided by Mental Health Services, with individual and family psychological therapies offered occasionally. Individual therapies may include CBT or psychodynamic interventions. To amend for the heterogeneity of TAU across centres, the type and extent of any treatment received will be protocolled at T1 and T2.

SUMMARY:
Auditory hallucinations (AH) are associated with distress and reduced functioning. Psychological interventions show some promising effects on psychopathology but have been less successful in reducing AH related distress, which patients report to be a priority. Research suggests that distress is associated with the hearer relating to AH in a passive and subordinate manner. A novel approach thus teaches assertive responses to AH through the use of experiential role-plays. A single centre pilot study in the United Kingdom evidenced a large effect of this approach on AH distress but independent multicentre studies are required to ascertain effectiveness across different settings. The planned feasibility trial aims to estimate the expected effect for a subsequent fully powered prospective, randomized, controlled, parallel-group, two-armed, multicentre, open trial set up to demonstrate that adding a Relating Module (RM) to Treatment as Usual (TAU) is superior to TAU alone. Feasibility questions relate to patient recruitment, therapist training and therapy monitoring in different types of psychological and psychiatric outpatient facilities.

DETAILED DESCRIPTION:
Auditory hallucinations (AH) are associated with distress and reduced functioning. Psychological interventions show some promising effects on psychopathology but have been less successful in reducing AH related distress, which patients report to be a priority. Research suggests that distress is associated with the hearer relating to AH in a passive and subordinate manner. A novel approach thus teaches assertive responses to AH through the use of experiential role-plays. A single centre pilot study in the United Kingdom evidenced a large effect of this approach on AH distress but independent multicentre studies are required to ascertain effectiveness across different settings. The planned feasibility trial aims to estimate the expected effect for a subsequent fully powered prospective, randomized, controlled, parallel-group, two-armed, multicentre, open trial set up to demonstrate that adding a Relating Module (RM) to Treatment as Usual (TAU) is superior to TAU alone. Feasibility questions relate to patient recruitment, therapist training and therapy monitoring in different types of psychological and psychiatric outpatient facilities. A total of 75 patients diagnosed with a schizophrenia spectrum disorder (ICD-10, F2) and persistent distressing AH will be recruited across 4 sites and receive either 16 50-minute sessions of RM plus TAU or TAU alone within a 5-months period. Assessments will take place at baseline, at 5 months (post-intervention) and at 9 months (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

Participants will;

1. have a diagnosis of a schizophrenia spectrum disorder (ICD-10, F2, confirmed by SCID-5)
2. patients will be reporting distressing AH for at least six months (to be beyond the startle and adjustment phase ) and score ≥ 3 on either item 8 or item 9 of the PSYRATS-AH;
3. be ≥ 16 years of age
4. be judged able to understand the full implications of their decision by the responsible psychiatrist or clinical psychologist.

Exclusion Criteria:

Participant must not:

1. have AH with a clear organic cause (e.g. brain disease or injury):
2. have exclusively hypnagogic or hypnopompic AH,
3. have a primary diagnosis of acute substance dependence (F1x.2)
4. have completed a course of CBT for psychotic symptoms during the past year within which distressing AH have been targeted
5. be currently participating, or be confirmed to participate in another interventional study in which they are receiving an intervention which utilizes psychological therapy ;
6. be non-German speaking to the degree that the participant is unable to fully understand and answer assessment questions or give informed consent;
7. be at immediate and serious risk to self or other.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
The Psychotic Symptom Rating Scales-AH-Distress factor score (PSYRATS-AH) | 9 months after baseline assessment
  Auditory hallucination associated distress. The distress factor score of the PSYRATS-AH is the primary outcome as this is what has been prioritized by patients and is relevant to functioning. Confirmatory analysis will be conducted based on the intent-to-treat population (ITT), defined on the basis of the ITT principle. The aim is to show that the intervention group is superior to the control meaning that the mean score at 9 months adjusted for the baseline value is lower in the intervention group than in the control group. Lower scores indicate less distress.

SECONDARY OUTCOMES:
Time Budget Measure | 5 and 9 months after baseline assessment
  Time that ist spent in social and vocational activities
EuroQuol Quality of Life Scale (EQ-5D-5L) | 5 and 9 months after baseline assessment
  Health-related quality of life
Columbia Suicide Severity Rating Scale (C-SSRS) | 5 and 9 months after baseline assessment
  Patients are interviewed about thoughts of wanting to complete suicide, active suicidal thoughts and intent to act on such thoughts (suicidal ideation, items 1-5) as well as about preparatory acts, aborted, interrupted or actual attempts (suicidal behaviour, 6-9). Completed suicide is rated on item 10. Scores on this scale range from 0 to 43 with higher scores indicating higher suicidal ideation
Number of rehospitalizations | 5 and 9 months after baseline assessment
  Number of hospitalizations after study enrollment
he Psychotic Symptom Rating Scales - PSYRATS-AH-Frequency | 5 and 9 months after baseline assessment
  Frequency of auditory hallucinations. Ranges from 0 to 4 with higher scores indicating higher frequency of auditory hallucinations
Patient Health Questionnaire-9 (PHQ-9) | 5 and 9 months after baseline assessment
  Self-report scale measuring depressive symptoms. Total score ranges from 0 to 21with higher scores indicating more severe depressive symptoms

OTHER OUTCOMES:
The Voice and You (VAY) | 5 and 9 months after baseline assessment
  To analyse whether the putative intervention effect is explicable by the changes in the processes targeted (improved relating to AH), two self-report scales will measure relating to AH. The VAY is a 29-item measure of interrelating between the hearer and their predominant voice (see above for a description of the development of this measure). Relating is measured across four scales; two concerning the hearer's perception of the relating of the voice-voice dominance and voice intrusiveness; and two concerning the relating of the hearer-hearer distance and hearer dependence. Each item is measured on a four-point scale (0-3). Higher scores indicate more negative relating.
Relating to Voices/Others Questionnaires (APPROVE) | 5 and 9 months after baseline assessment
  The APPROVE consists of two separate scales: A 46-item measure of relating to voices (Approve-Voices); and a 46-item measure of social relating (Approve-Social). The items were preceded by an introductory text inviting participants to "please select the answer that best reflects your typical response to [voices/other people] on the scale 0 (disagree completely) to 10 (agree completely). Where the item is not relevant to you then please select the not applicable (N/A) option". The following instruction - "When [voices/other people] are being difficult (e.g., treating me badly), I respond by: (...)" is presented before the list of the items (e.g., "Hearing what they are saying but also stating my own views").
Feasibility recruitment | through study completion, approximately two years after recruitment commenced
  Will count the number of patients referred within each site, number of self-referrals within each site, number of referred patients within each site found to be eligible, number and proportion of consenting and eligible participants who attend 5-month and 9 month assessment within each site
Feasibility completeness | through study completion, approximately 3 years after first participant has been randomized
  Will count the number and proportion of consenting participants within the RM condition who reach the point of therapy 'exposure' (attended at least 8 of 16 therapy sessions), percentage of complete of data sets
Therapist adherence | through study completion, an average of 4 weeks after baseline assessment
  All therapy sessions will be audio-recorded. For the first participant for each therapist, one recording from the early phase of therapy (sessions 1-6) and one recording from a later phase of therapy (sessions 7-14) will be randomly selected by the trial manager. The recordings will be translated, transcribed and sent to Dr Hayward for review. Therapist adherence to the treatment protocol will be assessed by Dr. Hayward who will assess two randomly selected recordings per therapist. Adherence will be rated using an adapted version of the Cognitive Therapy Scale for Psychosis (CTS-psy). Items F, G, and H have been adapted to include relating specific items in place of cognitive therapy (e.g. "Focus on the link between cognition and affect" was replaced with "focus on the effects of the patient engaging in different patterns of relating").
Safety monitoring | through study completion; 9 months after baseline assessment
  Will count the number of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tania M Lincoln, Prof. Dr., Principal Investigator — Universität Hamburg
Locations (5):
- Germany (5):
  - Universität Leipzig, Leipzig, Saxony
  - Klinik für Psychiatrie und Psychotherapie, Campus Benjamin Franklin Charité - Universitätsmedizin Berlin, Berlin
  - Jacobs University Bremen, Bremen
  - Psychotherapeutische Hoschschulambulanz Universität Hamburg, Hamburg
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No
only upon request

REFERENCES:
- [Result] Lincoln TM, Schlier B, Muller R, Hayward M, Fladung AK, Bergmann N, Boge K, Gallinat J, Mahlke C, Gonther U, Lang T, Exner C, Buchholz A, Stahlmann K, Zapf A, Rauch G, Pillny M. Reducing Distress from Auditory Verbal Hallucinations: A Multicenter, Parallel, Single-Blind, Randomized Controlled Feasibility Trial of Relating Therapy. Psychother Psychosom. 2024;93(5):328-339. doi: 10.1159/000539809. Epub 2024 Aug 21. PMID 39168112
- [Derived] Lincoln TM, Pillny M, Schlier B, Hayward M. RELATE-a randomised controlled feasibility trial of a Relating Therapy module for distressing auditory verbal hallucinations: a study protocol. BMJ Open. 2021 Jun 2;11(6):e046390. doi: 10.1136/bmjopen-2020-046390. PMID 34083338